CLINICAL TRIAL: NCT06806540
Title: The Frequency of Peripheral Arterial Disease in Patients with Deep Vein Thrombosis of the Lower Limbs
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: TVP-AOP
Record Dates: First submitted 2024-11-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-11

CONDITIONS: Thromboembolism; Peripheral Arterial Disease
Keywords: TVP; AOP
MeSH Terms: conditions — Thromboembolism; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of the study is to assess the frequency of Peripheral Arterial Disease (PAD) and cardiovascular risk factors in patients with unprovoked Deep Vein Thrombosis (DVT) of the lower limbs, comparing them with patients who have provoked DVT or cancer-related DVT. Additionally, the study aims to examine the association between the Ankle-Brachial Index (ABI) and Carotid Intima-Media Thickness (IMT) in the different patient groups.

This is an observational, spontaneous, monocentric, non-pharmacological study conducted on outpatient, non-hospitalized patients diagnosed with lower limb DVT, including both unprovoked and provoked DVT, as well as cancer-related DVT. The patients are followed at the Vascular Day Service of the SSD U.O. Angiology and Coagulation Disorders Unit at the Sant'Orsola Malpighi Polyclinic in Bologna. The study has a retrospective design for patients with DVT diagnosed between October 1, 2020, and the date of project approval, and a prospective design for patients diagnosed with DVT after this date. The study is expected to conclude by December 31, 2027.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the frequency of Peripheral Arterial Disease (PAD) and cardiovascular risk factors in patients with unprovoked Deep Vein Thrombosis (DVT) of the lower limbs, comparing them with patients with provoked DVT and cancer-related DVT. Additionally, the study aims to examine the association between Ankle-Brachial Index (ABI) and Carotid Intima-Media Thickness (IMT) in the different patient groups.

The study is an observational, spontaneous, monocentric, non-pharmacological study conducted on outpatients, non-hospitalized, who have been diagnosed with Deep Vein Thrombosis (DVT) of the lower limbs, either unprovoked or provoked, as well as cancer-related DVT. The patients are followed at the Vascular Day Service of the SSD U.O. Angiology and Coagulation Disorders at the Sant'Orsola Malpighi Hospital in Bologna. The study has a retrospective design for patients with DVT that occurred between October 1, 2020, and the project approval date, and a prospective design for patients who will experience DVT after this date, with the study scheduled to conclude by December 31, 2027.

The primary outcomes of the study are the frequency of PAD, defined as an ABI value below 0.90, in patients with unprovoked DVT compared to those with provoked DVT and cancer-related DVT; the measurement of carotid IMT and the presence of non-hemodynamic atherosclerotic plaques in patients with unprovoked DVT compared to the other groups; and finally, the analysis of the association between ABI, IMT measurements, and DVT. The secondary outcomes include the monitoring of recurrent thromboembolic events (DVT and/or Pulmonary Embolism - PE) and cardiovascular events (Acute Myocardial Infarction - AMI, Transient Ischemic Attack - TIA, stroke, peripheral ischemia), following patients according to standard clinical practice.

The study population includes all outpatients, non-hospitalized, who attend the Vascular Day Service of the SSD U.O. Angiology and Coagulation Disorders at the Sant'Orsola Malpighi Polyclinic in Bologna, with a diagnosis of Deep Vein Thrombosis (DVT) of the lower limbs, who underwent ultrasound evaluation for the diagnosis of deep venous thrombosis between October 1, 2020, and December 31, 2026 (study end date extended to December 31, 2023). At our center, patients are routinely managed following a clinical protocol that includes a clinical evaluation and an ultrasound examination in case of suspected DVT. If Pulmonary Embolism (PE) is suspected, a pulmonary CT angiography is performed. The pre-test clinical probability of DVT is assessed using the Wells score, with the following values:

* < 1: low probability of DVT
* 1-2: moderate probability of DVT
* > 2: high probability of DVT

Patients are then subjected to real-time compression ultrasound (B-mode) and color Doppler ultrasound of the entire deep venous system, using a high-resolution linear probe (12-5 MHz) with a Logiq5 machine, General Electrics. The diagnosis of DVT is confirmed when the absence of compressibility in the deep venous axis is found, along with the absence of venous flow on distal compression. The ultrasound (CUS) results are recorded in a standardized data collection form, also indicating the anatomical location of the DVT (proximal, distal, and affected venous segments).

For analytical purposes, patients will be divided into three groups based on the nature of the deep vein thrombosis event:

* Group 1: Unprovoked DVT
* Group 2: Provoked DVT
* Group 3: Cancer-related DVT

Provoked DVT will be considered as such when associated with: Surgery; Trauma; Lower limb immobilization; Long air travel; Use of estrogen-progestin medications; Hospitalization with bed rest > 3 days in the previous three months.

All patients diagnosed with DVT will be evaluated for the presence of Peripheral Arterial Disease (PAD), with diagnosis based on the presence of at least one of the following criteria:

* Previous arterial revascularization surgery on a limb,
* Previous limb amputation due to arterial disease,
* Previous carotid revascularization or carotid stenosis ≥ 50%,
* Instrumental findings of: ABI ≤ 0.9; Carotid IMT; Femoral IMT.

The Ankle-Brachial Index (ABI) is a simple, non-invasive clinical test used to diagnose peripheral artery disease. It is calculated as the ratio of distal peripheral arterial pressure (measured in both anterior and posterior tibial arteries) to brachial arterial pressure. The ABI values are interpreted as follows: • ABI ≥ 1.4: incompressible artery

* ABI between 1 and 1.3: normal
* ABI ≤ 0.9: presence of peripheral artery disease: Moderate, if ABI between 0.4 and 0.9; Severe, if ABI < 0.4.

Intima-Media Thickness (IMT) of the carotid or femoral arterial wall is used as a marker for early atherosclerotic changes. IMT is measured as the distance between the inner hyperechoic line of the vascular wall (blood-intima interface) and the outer hyperechoic line (media-adventitia interface). IMT values are classified as follows:

* IMT < 0.8 mm: normal
* IMT between 0.8 and 1.4 mm: medium-intimal thickening
* IMT ≥ 1.5 mm: atheromatous plaque

ABI and IMT values will be recorded in a standardized data collection form.

Inclusion criteria for the study sample include: Age ≥ 18 years; Diagnosis of unprovoked, provoked, or cancer-related DVT; Diagnosis of DVT in the lower limbs (either proximal or distal), with compression ultrasound within 6 months of diagnosis; Ability to provide informed consent.

Exclusion criteria include: Diagnosis of upper limb DVT or DVT in other locations, unless concurrent with lower limb DVT; Diagnosis of Superficial Venous Thrombosis (SVT), unless concurrent with lower limb DVT; Diagnosis of DVT associated with Central Venous Catheters (CVC); Presence of epithelomas/basal cell carcinomas, as these are associated with a low risk of DVT.

The study aims to provide a deeper understanding of the relationship between DVT, PAD, and cardiovascular risk factors, in order to improve the clinical management of patients with deep vein thrombosis and cardiovascular comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of unprovoked, provoked, or cancer-related DVT
* Diagnosis of DVT in the lower limbs, both proximal and distal, subjected to compression ultrasound within 6 months of diagnosis
* Ability to provide informed consent

Exclusion Criteria:

* Diagnosis of upper limb DVT or DVT in other locations, if not concurrent with lower limb DVT
* Diagnosis of superficial venous thrombosis (SVT), if not concurrent with lower limb DVT
* Diagnosis of DVT associated with central venous catheters (CVC)
* Presence of epithelial or basal cell carcinomas, as they are associated with a low risk of deep vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All outpatients, not admitted to the hospital, attending the Vascular Day Service of the SSD U.O. Angiology and Coagulation Disorders Unit at the Sant'Orsola Malpighi Polyclinic in Bologna will be evaluated from 01/10/2020 to 31/12/2026.
  At our center, these patients are typically managed according to the standard care pathway, which includes a clinical evaluation and an ultrasound examination in case of suspected deep vein thrombosis (pulmonary CT angiography in the case of suspected pulmonary embolism).
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of POA (Peripheral Obliterative Arteriopathy) | Through study completion, an average of 1 year
  Among the first-line non-invasive tests useful both for the diagnosis and surveillance of POA and for defining cardiovascular risk is the ABI (Ankle Brachial Index). The ABI is calculated as the ratio between the systolic pressure measured at the level of the posterior tibial artery (ankle) (or at the level of the pedal artery) of each limb and the systolic pressure measured bilaterally at the brachial artery (upper arm). The highest pressure value measured at each site is used for the calculation. The most commonly used method for measuring pressure involves the use of an 8 MHz CW Doppler probe. The primary outcome will be to assess the frequency of AOP defined by an ABI < 0.90 in patients with unprovoked DVT compared to patients with provoked DVT and cancer-associated DVT.
Assess the presence of atherosclerotic plaques and the IMT (Intima-Media Thickness)of the common carotid artery | Through study completion, an average of 1 year
  Arterial color Doppler ultrasound is among the first-line non-invasive tests useful both for the diagnosis and surveillance of POA as well as for defining cardiovascular risk. In particular, color Doppler of the supra-aortic trunks allows the evaluation of atherosclerotic plaques and the IMT of the common carotid artery, which is widely used as a surrogate marker of diffuse atherosclerotic disease. Therefore, IMT and/or non-hemodynamic atherosclerotic plaques are assessed in patients with unprovoked DVT compared to patients with provoked DVT and cancer-associated DVT
Evaluate the correlation between ABI, IMT measurements, and DVT | Through study completion, an average of 1 year
  The aim is to evaluate the correlation between ABI, IMT measurements, and DVT, as some studies have shown a significant association between them, but the data in the literature are limited

SECONDARY OUTCOMES:
Monitoring Thromboembolic Recurrence and Cardiovascular Events in Patients Following Standard Clinical Care | Through study completion, an average of 1 year
  Patients will be followed according to standard clinical practice, with monitoring of thromboembolic recurrence events (DVT and/or PE) and cardiovascular events (MI, TIA, stroke, peripheral ischemia).

CONTACTS AND LOCATIONS:
Overall Officials: Benilde Cosmi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azianda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy